CLINICAL TRIAL: NCT07333352
Title: Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of A 24-Valent Pneumococcal Polysaccharide Conjugate Vaccine (RZ700) in Infants and Young Children Aged 2 Months (Minimum 6 Weeks) to 71 Months
Brief Title: PCV24 Clinical Trial in Infants and Young Children Aged 2 Months (Minimum 6 Weeks) to 71 Months
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Reinovax Biologics Co.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RNCVCT7B002
Record Dates: First submitted 2025-12-01; First posted 2026-01-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pneumococcal Infectious Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort I :2 months (minimum 6 weeks）of age. (Experimental): Subjects aged 2 months (minimum 6 weeks) will receive the experimental vaccine or comparator control vaccine according to 0, 2, and 4-month immunization schedule, followed by a booster dose at 12-15 months of age.
  Interventions: Biological: 24-Valent Pneumococcal Polysaccharide Conjugate Vaccine (RZ700); Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine (Prevnar 13)
- Cohort II : 7~23 months of age. (Experimental): Subjects aged 7-11 months will receive the experimental vaccine or comparator control vaccine according to the 0 and 2-month immunization schedule. A booster dose will be administered at 12-15 months of age. Accprdingly, subjects aged 12-23 months will receive the experimental vaccine or comparator control vaccine according to the 0 and 2-month immunization schedule.
  Interventions: Biological: 24-Valent Pneumococcal Polysaccharide Conjugate Vaccine (RZ700); Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine (Prevnar 13)
- Cohort III : 24~71 months of age. (Experimental): Subjects aged 24-71 months will receive a single intramuscular injection of the experimental vaccine or comparator control vaccineon the day of enrollment.
  Interventions: Biological: 24-Valent Pneumococcal Polysaccharide Conjugate Vaccine (RZ700); Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine (Prevnar 13)

INTERVENTIONS:
Biological: 24-Valent Pneumococcal Polysaccharide Conjugate Vaccine (RZ700) — 24-Valent Pneumococcal Polysaccharide Conjugate Vaccine (RZ700) consisting of polysaccahrides from 24 pneumococcal serotypes: 1, 2, 3, 4, 5, 6A, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F conjugated two carrier proteins. Each dose contains 0.5 ml vaccine in a prefilled syringe.
Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine (Prevnar 13) — 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine (Prevnar 13) consisting of plosaccharides from 13 pneumococcal serotypes: 1, , 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F conjugated CRM197. Each dose contains 0.5 ml vaccine in a prefilled syringe.

SUMMARY:
The Phase II clinical trial of the 24-valent pneumococcal polysaccharide conjugate vaccine (RZ700) will be carried out in infants and young children aged 2 months (minimum 6 weeks) to 71 months. The purpose of this study is to evaluate the immunogenicity and safety of the 24-valent pneumococcal polysaccharide conjugate vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 2 months (minimum 6 weeks) and 7-71 months, whose guardians can provide valid identification documents for both the subjects and themselves, as well as proof of their guardianship relationship.
* The guardians of the subjects voluntarily agree to their participation in this trial, sign the Informed Consent Form (ICF), and are willing to comply with all requirements of this clinical trial protocol.
* The guardians of the subjects have the ability to understand the trial procedures (non-illiterate).

Exclusion Criteria:

* Subjects who have received any type of pneumococcal vaccine prior to enrollment, plan to receive a pneumococcal vaccine during the trial, or have a history of invasive diseases caused by Streptococcus pneumoniae (confirmed by any clinical, serological, or microbiological method).
* Subjects with abnormal physical examination results that are deemed clinically significant by a clinician.
* Subjects with suspected or confirmed fever (axillary temperature ≥ 37.5℃) within 3 days prior to enrollment; or those with an axillary temperature ≥ 37.5℃ on the day before the first dose of vaccination.
* Subjects with a history of acute illness, acute exacerbation of chronic illness, systemic use of antibiotics or antiviral drugs within 3 days prior to the first dose of vaccination; or those who have taken antipyretic, analgesic, or antiallergic drugs (e.g., acetaminophen, ibuprofen, loratadine, cetirizine, etc.) within 3 days prior to the first dose of vaccination.
* Subjects with a history of allergy to any component of the study vaccine, any vaccine containing tetanus toxoid, or a previous history of severe allergy to any vaccine or drug (including but not limited to anaphylactic shock, allergic laryngeal edema, allergic purpura, immune thrombocytopenic purpura, local allergic necrotizing reaction, dyspnea, angioedema, etc.); or a previous history of the aforementioned severe adverse reactions following the use of any vaccine or drug.
* Subjects who have received inactivated vaccines, subunit vaccines, or recombinant vaccines within 7 days prior to enrollment; or live attenuated vaccines, adenovirus vector vaccines, etc., within 14 days prior to enrollment.
* Subjects who have received any other investigational drugs within 3 months prior to enrollment or plan to use them during the trial; those who have received whole blood, plasma, or blood products (e.g., immunoglobulin therapy) within 3 months prior to enrollment or plan to receive such treatments during the trial.
* Subjects with a history of thrombocytopenia, idiopathic thrombocytopenic purpura, or other coagulation disorders diagnosed by a hospital; or a history of receiving anticoagulant therapy.
* Subjects with a known current or past history of infectious diseases diagnosed by a hospital, such as active tuberculosis, hepatitis B, hepatitis C, HIV infection, etc.
* Subjects with known or suspected severe chronic diseases (e.g., liver and kidney diseases, malignant tumors, infectious or allergic skin diseases, hemolytic uremic syndrome); or those whose condition is in the progressive stage and cannot be stably controlled.
* Infants aged 2 months (minimum 6 weeks) and 7-11 months with abnormal birth weight (<2500g), abnormal gestational age (<37 weeks or >42 weeks), abnormal delivery (dystocia, instrumental delivery), or a history of asphyxia or neuroorganic damage.
* Infants aged 2 months (minimum 6 weeks) and 7-11 months with severe eczema or severe jaundice (grade 3 or above).
* Subjects with severe congenital malformations, developmental disorders, genetic defects, severe malnutrition, or severe chronic diseases (e.g., tetralogy of Fallot, tricuspid atresia, Down syndrome, sickle cell anemia, etc.).
* Subjects with neurological diseases or neurodevelopmental disorders (e.g., febrile convulsions, epilepsy, encephalopathy, focal neurological deficits, encephalomyelitis or transverse myelitis, Guillain-Barré syndrome); or a history of mental illness in the subjects themselves or their biological parents.
* Subjects with a history of congenital or acquired immunodeficiency, immunosuppression, or autoimmune diseases; or those who have received immunomodulatory therapy within 6 months (e.g., immunosuppressive doses of glucocorticoids [dosage reference: equivalent to prednisone ≥0.5mg/kg/day for more than 2 weeks], monoclonal antibodies, thymopeptides, interferons, etc.); or plan to receive such treatments from enrollment to 30 days after the last dose of vaccination. Topical medications (e.g., ointments, eye drops, inhalants, or nasal sprays) are permitted.
* Subjects with asplenia, functional asplenia, or asplenia/resplenectomy caused by any condition.
* Subjects whose guardians may be unable to comply with trial procedures, adhere to agreements, plan to permanently relocate from the region before the trial is completed, or be away from the local area for a long time during scheduled visits.
* Researchers believe that the subject has any other factors that make them unsuitable for participating in the clinical trial, such that continued participation cannot ensure the subject's maximum benefit.

Ages: 6 Weeks to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with the pneumococcal serotype-specific IgG antibody concentration ≥0.35 μg/ml. | 30 days post the primary and booster immunization.
  Proportion of subjects with the pneumococcal serotype-specific IgG antibody concentration ≥0.35 μg/ml.

SECONDARY OUTCOMES:
The proportion of subjects with serum IgG antibody concentration ≥1.0 μg/ml against 24 serotypes of Streptococcus pneumoniae. | 30 days after completion of the primary immunization schedule
  The proportion of subjects aged 2 months (minimum 6 weeks old) and 7~71 months old with serum IgG antibody concentration ≥1.0 μg/ml against 24 serotypes of Streptococcus pneumoniae.
Pneumococcal serotype-specific IgG antibody geometric mean fold rise (GMFR) against 24 serotypes post immunization compared with pre-immunization. | 30 days after completion of the primary immunization schedule.
  Pneumococcal serotype-specific IgG antibody geometric mean fold rise (GMFR) against 24 serotypes in subjects aged 2 months (minimum 6 weeks old) and 7~71 months old compared with pre-immunization.
Pneumococcal serotype-specific IgG antibody geometric mean concentration (GMC) . | 30 days after completion of the primary immunization schedule
  Pneumococcal serotype-specific IgG antibody geometric mean concentration (GMC) for each serotype (1, 2, 3, 4, 5, 6A, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F) in subjects aged 2 months (minimum 6 weeks old) and 7~71 months old at 30 days after completion of the primary immunization.
The proportion of subjects with serum IgG antibody concentration ≥1.0 μg/ml against 24 serotypes of Streptococcus pneumoniae. | 30 days after completion of the booster immunization schedule
  The proportion of subjects aged 2 months (minimum 6 weeks old) and 7~11 months old with serum IgG antibody concentration ≥1.0 μg/ml against 24 serotypes of Streptococcus pneumoniae.
The proportion of subjects with serum MOPA titer ≥1:8 against Streptococcus pneumoniae. | 30 days after vaccination
  The proportion of subjects in the MOPA testing subgroup aged 24~71 months with serum MOPA titer ≥1:8 against Streptococcus pneumoniae.
Geometric Mean Titer (GMT) of pneumococcal serotype-specific MOPA antibodies in serum. | 30 days after vaccination
  Pneumococcal serotype-specific MOPA geometric mean titer (GMT) in serum of subjects aged 24~71 months in the MOPA testing subgroup.
Pneumococcal serotype-specific MOPA geometric mean titer fold rise (GMFR) in serum. | 30 days after vaccination
  Pneumococcal serotype-specific MOPA geometric mean titer fold rise (GMFR) in serum of subjects aged 24~71 months in the MOPA testing subgroup.
Incidence rate of all adverse events (AEs). | Within 30 days after each dose of vaccination
  Incidence rate of all adverse events (AEs) within 30 minutes, 7 days, and 30 days after each dose of vaccination in each age group.
Occurrence of serious adverse events (SAEs) and adverse events of special interest (AESIs). | From the first dose of vaccination to 6 months after completion of the full vaccination course
  12~71 months old: Occurrence of serious adverse events (SAEs) and adverse events of special interest (AESIs).
Occurrence of serious adverse events (SAEs) and adverse events of special interest (AESIs). | From the first dose of the primary immunization course to 6 months after completion of the booster immunization
  2 months old (minimum 6 weeks old)and 7 to 11 months old: Occurrence of serious adverse events (SAEs) and adverse events of special interest (AESIs).

CONTACTS AND LOCATIONS:
Overall Officials: Yunong Zhang, Master, Principal Investigator — Shanxi Province Center for Disease Control and Prevention
Locations (7):
- China (7):
  - Luzhou District Center for Disease Control and Prevention, Changzhi, Shanxi
  - Qinxian County Center for Disease Control and Prevention, Changzhi, Shanxi
  - Kuangqu District Center for Disease Control and Prevention of Yangquan City, Yangquan, Shanxi
  - Xinjiang County Center for Disease Control and Prevention, Yuncheng, Shanxi
  - Jishan County Center for Disease Control and Prevention, Yuncheng, Shanxi
  - Yongji City Center for Disease Control and Prevention, Yuncheng, Shanxi
  - Shangdang District Center for Disease Control and Prevention of Changzhi City, Yuncheng, Shanxi

IPD SHARING:
Plan to Share IPD: No